CLINICAL TRIAL: NCT04147819
Title: A Phase 1 Open-label, First-in-human, Multi-center Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Anti-tumor Activity of Thorium-227 Labeled Antibody-chelator Conjugate BAY2701439, in Participants With Advanced HER2-expressing Tumors
Brief Title: A First in Human Study of BAY2701439 to Look at Safety, How the Body Absorbs, Distributes and Excretes the Drug, and How Well the Drug Works in Participants With Advanced Cancer Expressing the HER2 Protein
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 19829; 2019-001741-40 (EudraCT Number)
Record Dates: First submitted 2019-10-25; First posted 2019-11-01 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Cancers With HER2 Expression
Keywords: Human epidermal growth factor receptor 2(HER2); Targeted alpha therapy; Thorium-227; HER2 low; HER2-low; HER2 positive; HER2-positive; HER2 expressing; HER2-expressing; Breast cancer; Gastric cancer
MeSH Terms: conditions — Breast Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose escalation of BAY2701439 (Experimental): The target population consists of participants with advanced HER2-expressing/amplified breast, gastric or gastroesophageal cancer.
  Interventions: Drug: BAY2701439
- HER2 overexpressing breast cancer (Experimental): Dose expansion of BAY2701439
  Interventions: Drug: BAY2701439
- HER2 low expressing breast cancer (Experimental): Dose expansion of BAY2701439
  Interventions: Drug: BAY2701439
- Other HER2 overexpressing advanced carcinomas (Experimental): Dose expansion of BAY2701439
  Interventions: Drug: BAY2701439

INTERVENTIONS:
Drug: BAY2701439 — Intravenous (IV) injection on Day 1 of each cycle.The duration of each cycle will be 6 weeks (42 days).
Drug: BAY2701439 — Intravenous (IV) injection on Day 1 of each cycle and 1 hour before the start of administration of BAY2701439. The duration of each cycle will be 6 weeks (42 days).

SUMMARY:
In this study, researchers want to learn about the safety of drug BAY2701439 and how well the drug works in patients with advanced cancer that has the protein HER2 (Human Epidermal growth factor Receptor 2) and cannot be cured by currently available treatment options. The study will include patients with HER2 expressing breast, gastric (stomach) or gastroesophageal (stomach and esophagus) cancer, as well as other cancers that have HER2. Researchers want to find the best dose of BAY2701439 for patients and look at the way the body absorbs, distributes and excretes the drug.

The study drug is a type of therapy called a 'targeted alpha therapy' which uses an antibody to deliver a radioactive particle to cancer cells. BAY2701439 contains thorium-227 which emits radiation (a lot of energy that moves from one place to another with damaging effects). The thorium-227 in the drug is attached to an 'antibody' (large protein) that specifically binds to HER2 on the cancer cells and will emit its radiation in the form of alpha particles. The alpha particles are expected to damage the tumor cells and cause them to die, but spare surrounding tissue as alpha particles travel only very short distances in the body. This is the first study in humans for drug BAY2701439. Patients participating in this study will receive the drug by injection every 6 weeks a maximum 6 times. Observation after treatment last up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants at least 18 years of age on the day of signing informed consent.
* Participants must meet the study phase-specific disease requirements:

Dose escalation:

Pathologically documented, HER2-expressing (IHC3+, 2+, or 1+ and/or ISH+), unresectable locally advanced or metastatic gastric, gastroesophageal, or breast cancer that has relapsed after standard treatment options, or for which no standard treatment is available. Participants with gastric or gastroesophageal cancer must not have had prior definitive radiotherapy. Participants in the dose escalation cohorts must have evaluable disease by RECIST 1.1, assessed by local imaging.

- Dose expansion: Group A: Pathologically documented unresectable, locally advanced or metastatic breast cancer with HER2 overexpression or amplification (IHC3+ or IHC2+/ISH+) that has relapsed that has relapsed after standard treatment options, or for which no standard treatment is available.

Group B: Pathologically documented unresectable locally advanced or metastatic breast cancer with HER2 low expression (IHC2+/ISH-, IHC1+/ISH-, or IHC1+/ISH untested) that has relapsed after standard treatment options, or for which no standard treatment is available.

Group C: Pathologically documented, unresectable locally advanced or metastatic carcinomas other than breast cancer with HER2 overexpression or amplification/mutation (IHC3+ or IHC2+/ISH+), that has relapsed after standard treatment options or for which no standard treatment is available.

Participants in the dose expansion cohorts must have measurable disease by RECIST 1.1, assessed by local imaging.

* Availability of fresh or archival tumor samples - archival tumor samples obtained after disease progression on the most recent anti-cancer treatment may be accepted; those obtained prior to the last anti-cancer treatment may be accepted, upon agreement between the Sponsor and the Investigator.
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1.
* Life expectancy of at least 6 months, as estimated by the Investigator.
* Adequate bone marrow, hepatic, and renal function, as assessed by the following laboratory requirements, to be conducted within 28 days before start of BAY2701439 administration:

  * Hemoglobin ≥ 9.0 g/dL
  * Absolute neutrophil count (ANC) ≥ 1500/mm*3
  * Platelet count ≥ 100,000/mm*3
  * Total bilirubin ≤ 1.5 X the upper limit of normal (ULN), except if confirmed history of Gilbert's disease
  * Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) ˂ 2.5 x ULN (≤ 5 x ULN for participants with liver involvement)
  * Participants on a stable dose of anti-coagulation therapy will be allowed to participate if they have no sign of bleeding or clotting, and Prothrombin time/International normalized ratio (PT/INR) and aPTT test results are compatible with the acceptable benefit-risk ratio at the Investigator's discretion
  * Serum creatinine ≤ 1.5 x ULN and glomerular filtration rate (GFR)≥ 45 mL/min/1.73 m*2, according to the Modified Diet in Renal Disease (MDRD)abbreviated formula.
* A negative serum pregnancy test in women of childbearing potential (WOCBP) performed within 7 days before the start of BAY2701439 administration. Women and men of reproductive potential must agree to use highly effective methods of contraception, when sexually active, during the time period between signing the informed consent form until at least 6 months after the last administration of BAY2701439.
* Male and/or female who meet the requirements for contraception and breastfeeding as follows:

Male participants: A male participant must agree to use highly effective contraception during the intervention period and for at least 6 months after intervention and refrain from donating sperm during this period.

Female participants: A female participant is eligible to participate if she is not pregnant (confirmed by a negative serum pregnancy test within 7 days of first study treatment), not breastfeeding, or is not a woman of childbearing potential.

Women of childbearing potential (WOCBP) must agree to use highly effective contraception during the intervention period and for at least 6 months after the last dose of study treatment.

Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

- Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol

Exclusion Criteria:

* Impaired cardiac function or clinically significant cardiac disease (i.e. congestive heart failure (CHF) New York Heart Association (NYHA) Class II, III or IV).
* Left ventricular ejection fraction (LVEF) < 50% (as measured at screening by echocardiogram).
* History or concurrent condition of interstitial lung disease/pneumonitis or severely impaired pulmonary function.
* Participants known to be affected by genetic defects linked to radiation hypersensitivity, such as ataxia-telangiectasia (A-T; Online Mendelian Inheritance in Man [OMIM] #208900) and A-T-like disorder (meiotic recombination 11 homolog [MRE11]), Nijmegen breakage syndrome (OMIM #251260) and Nijmegen breakage Syndrome-like disorder (RAD50), Fanconi anemia (OMIM #227650), DNA ligase IV deficiency (OMIM #606593), RIDDLE syndrome (RNF168), radiosensitive severe combined immunodeficiency (RS-SCID), DNA-PK radiosensitive combined immunodeficiency (DNA-PK-RS-SCID), Cornelia de Lange syndrome.
* History of Myelodysplastic syndrome (MDS)/treatment-related acute myeloid leukemia (t-AML) or with features suggestive of MDS/AML.
* Infections of Common terminology criteria for adverse events (CTCAE) version 5.0 Grade 2 not responding to therapy or active clinically serious infections of CTCAE Grade >2.
* History of hypersensitivity or severe infusion related reaction to any Trastuzumab-containing drug (e.g. trastuzumab, T-DM1) or any other ingredients contained in BAY2701439.
* Chemotherapy, experimental cancer therapy, biologic therapy or immunotherapy within 4 weeks before start of BAY2701439 administration. Start of study treatment is allowed in shorter timeframes provided 5 half-lives of the prior drug(s) have elapsed before the start of BAY2701439 administration. Previous high-dose chemotherapy needing hematopoietic-stem-cell-rescue is prohibited.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-07-02 (Actual); Primary Completion 2023-08-21 (Actual); Study Completion 2023-09-26 (Actual)

PRIMARY OUTCOMES:
Dose escalation: Incidence of TEAEs including TESAEs | After first administration of study intervention up to 42 days after the last dose of study intervention
  TEAE: Treatment-emergent adverse event TESAE: Treatment-emergent serious adverse event
Dose escalation: Severity of TEAEs including TESAEs | After first administration of study intervention up to 42 days after the last dose of study intervention
Dose escalation: Frequency of DLTs at each dose level | Up to 42 days after first administration of study intervention on cycle 1 (42 days) day 1
  DLT:Dose limiting toxicity
Dose expansion: ORR by RECIST 1.1 based on Investigator review | Up to 12 months after End of treatment
  ORR: Objective response rate
Dose expansion: Frequency of TEAEs | After first administration of study intervention up to 42 days after the last dose of study intervention
Dose expansion: Severity of TEAEs | After first administration of study intervention up to 42 days after the last dose of study intervention

SECONDARY OUTCOMES:
Dose escalation: Recommended dose level(s) of BAY2701439 for the dose expansion cohorts | Maximum 6 cycles (each cycle is 42 days)
  The dose level(s) recommended for the dose expansion cohorts will be defined after evaluation of incidence and severity of TEAEs, PK, and ORR by RECIST 1.1, collected in the cycles of treatment during the dose escalation part of the study.
Dose escalation: Recommended treatment schedule of BAY2701439 for the dose expansion cohorts | Maximum 6 cycles (each cycle is 42 days)
  The treatment schedule recommended for the dose expansion cohorts will be defined after evaluation of incidence and severity of TEAEs, PK, and ORR by RECIST 1.1, collected in the cycles of treatment during the dose escalation part of the study.
Dose expansion: Recommended dose for further clinical development of BAY2701439 | Maximum 6 cycles (each cycle is 42 days)
  The dose recommended for further clinical development will be defined after evaluation of incidence and severity of TEAEs, PK, and ORR by RECIST 1.1, collected in the cycles of treatment during the dose escalation and expansion parts of the study.
Cmax of thorium-227 | Cycle 1 (42 days)
  Cmax: Maximum observed exposure
Cmax of radium-223 | Cycle 1 (42 days)
  Cmax: Maximum observed exposure
Cmax of total antibody | Cycle 1 (42 days)
  Cmax: Maximum observed exposure
AUC(0-42 days) of thorium-227 | Cycle 1 (42 days)
  AUC: Area under the curve
AUC(0-42 days) of radium-223 | Cycle 1 (42 days)
  AUC: Area under the curve
AUC(0-42 days) of total antibody | Cycle 1 (42 days)
  AUC: Area under the curve

CONTACTS AND LOCATIONS:
Locations (6):
- United States (4):
  - Johns Hopkins Hospital/Health System, Baltimore, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- United Kingdom (2):
  - Southampton General Hospital, Southampton, Hampshire
  - Royal Marsden NHS Trust (Surrey), Sutton, Surrey

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- [Derived] Anderson PM, Subbiah V, Trucco MM. Current and future targeted alpha particle therapies for osteosarcoma: Radium-223, actinium-225, and thorium-227. Front Med (Lausanne). 2022 Nov 15;9:1030094. doi: 10.3389/fmed.2022.1030094. eCollection 2022. PMID 36457575
- See also: Click here to find further information and, after study completion, the study results according to Bayer's transparency standards. — https://clinicaltrials.bayer.com/study/19829